CLINICAL TRIAL: NCT05209152
Title: A Phase 1 Study of AMG 176 as Monotherapy and in Combination With Azacitidine in Higher-Risk Myelodysplastic Syndrome and Chronic Myelomonocytic Leukemia
Brief Title: AMG 176 With Azacitidine in Subjects With Myelodysplastic Syndrome /Chronic Myelomonocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision, unrelated to safety
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20200392
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Higher Risk Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
Keywords: Higher Risk Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — tapotoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A - AMG 176 Monotherapy (Dose Exploration) (Experimental): Two dose levels of AMG 176 will be tested in Part 1A to find the optimal biological dose/minimum safe biologically effective dose (OBD/MSBED).
  Interventions: Drug: AMG 176
- Part 1B - AMG 176 and Azacitidine Combination Therapy (Dose Exploration) (Experimental): After the OBD is found in Part 1A, two dose levels of AMG 176 in combination with azacitidine will be tested in Part 1B to find the OBD/MSBED.
  Interventions: Drug: AMG 176; Drug: Azacitidine
- Part 2 - AMG 176 and Azacitidine Combination Therapy (Dose Expansion) (Experimental): After the completion of Part 1, the Part 2 dose expansion phase will begin at the OBD/MSBED identified in Part 1.
  Venetoclax-naïve and venetoclax-exposed R/R HR-MDS participants after HMA failure will be enrolled along with participants with newly diagnosed HR-MDS/CMML.
  Interventions: Drug: AMG 176; Drug: Azacitidine

INTERVENTIONS:
Drug: AMG 176 — Administered as an intravenous (IV) infusion.
Drug: Azacitidine — Administered as an IV infusion or subcutaneous (SC) injection.
  Arms: Part 1B - AMG 176 and Azacitidine Combination Therapy (Dose Exploration); Part 2 - AMG 176 and Azacitidine Combination Therapy (Dose Expansion)

SUMMARY:
The main objective is to assess the safety, tolerability, and efficacy of AMG 176 as monotherapy and in combination with the 7-day regimen of azacitidine for the treatment of Higher-Risk Myelodysplastic Syndrome and Chronic Myelomonocytic Leukemia (HR-MDS/CMML).

DETAILED DESCRIPTION:
This study is a Phase 1 clinical trial designed to assess the safety, tolerability, and efficacy of AMG 176 as monotherapy and in combination with the 7-day regimen of azacitidine for the treatment of HR-MDS/CMML. Participants will be treated with intravenous (IV) AMG 176 and IV or subcutaneous (SC) azacitidine.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* For Part 1, participants have R/R MDS post-HMA failure, defined as prior receipt of 4 cycles of HMA therapy (including but not limited to decitabine, azacitidine, investigational HMAs such as SGI-110, and oral HMAs such as oral decitabine and cedazuridine [ASTX727] and oral azacitidine [CC-486]) with failure to attain a response or progression of disease or relapse at any time after prior response to HMA therapy

  a. Note: participants with HR-CMML (CMML-1 or 2 by World Health Organization [WHO]) are eligible. Hydroxyurea administration will be allowed on the study to lower the white cell count to <= 10 000/μL prior to the initiation of therapy
* For Part 2, participants will be divided into 2 cohorts:

  1. HMA Failure Cohort: participants with R/R MDS post-HMA failure. Participants who have previously received venetoclax are eligible and will be stratified accordingly in the HMA failure cohort;
  2. Newly Diagnosed Cohort: Participants with treatment-naïve newly diagnosed HR-MDS (revised International Prognostic Scoring System [IPSS-R] score >3.5) are eligible for enrollment only after all prior cohorts have been completed. Hydroxyurea administration will be allowed on the study to lower the white cell count to <= 10 000/μL prior to the initiation of therapy. Participants with HR-CMML (CMML-1 or 2 by WHO) are eligible

Exclusion Criteria:

* Participants with newly diagnosed MDS with Revised International Prognostic Scoring System (IPSS-R) lower-risk category (IPSS-R score < 3.5)
* Participants with CMML-0 by WHO
* History of other malignancy within the past 2 years prior to enrollment (with some exceptions as listed in full list of criteria)
* Excluded prior and/or concomitant therapies as listed in the full list of criteria
* Participants who are fit and deemed eligible by the investigator for intensive salvage therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7 participants with higher risk myelodysplastic syndromes (MDS) and chronic myelomonocytic leukemia were enrolled at a single study center in the United States from November 2022 and the last participant's last visit was in December 2023.
Pre-assignment Details: The study was planned to be conducted in 3 parts and was discontinued early after the completion of Part 1A (dose exploration). Part 1B (dose escalation/de-escalation) and Part 3 (dose expansion) were not conducted and did not enroll any participants. Dose level 1 is a low dose and Dose level 2 is a high dose.
Groups:
- Part 1A Dose Exploration: AMG 176 Dose Level 1: Participants received intravenous (IV) AMG 176 at dose level 1 once a week in 28-day cycles. Treatment was planned until disease progression or unacceptable toxicity.
- Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2: Participants received IV AMG 176 at dose level 1 on cycle 1 day 1 and then dose level 2 from cycle 1 day 8 and once a week thereafter (each cycle = 28 days). Treatment was planned until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Sponsor decision | 1 | 2
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1A Dose Exploration: AMG 176 Dose Level 1: Participants received IV AMG 176 at dose level 1 once a week in 28-day cycles. Treatment was planned until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2 | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 6
  Black or African American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: DLTs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and included the below if considered by the investigator to be related to AMG 176: Grade 3 or higher non-hematological or a Grade 4 hematologic adverse event (AE) during the DLT observation period in Part 1.
  CTCAE Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, and Grade 5 results in death.
Time Frame: Day 1 to day 28 of cycle 1 (each cycle was 28 days)
Population: DLT-evaluable participants were those who experienced a DLT during the DLT evaluation period or if they received 75% of the planned doses of AMG 176 and completed the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical trial participants. TEAEs were any AE that started on or after receiving the first dose of investigational product and up to 28 days after the last dose of investigational product or the end of study date, whichever is earlier. Treatment-related TEAEs were those considered possibly related to study treatment by the investigator. Any clinically significant changes in electrocardiograms, vital signs, and clinical laboratory tests were recorded as TEAEs. A serious TEAE resulted in death, was immediately life threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Time Frame: Day 1 cycle 1 to 30 days after the last dose of AMG 176 or end of study, whichever occurred earlier (cycle length = 28 days). Median treatment duration was 2.7 months
Population: The full analysis set included all enrolled participants who received at least 1 dose of AMG 176.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
Participants
  Any TEAE | 4 | 3
  Any serious TEAE | 3 | 2

3. Secondary Outcome: Number of Participants With a Response According to the Uniform Response Criteria for MDS/Myeloproliferative Neoplasm (MPN)
Description: A responder was assessed as having complete remission (CR) or partial remission (PR). Non-responders had stable disease, progressive disease or were not evaluable.
  CR: ≤ 5% myeloblasts with normal maturation of all cell lines and return to normal cellularity; osteomyelofibrosis was absent or equal to mild reticulin fibrosis; resolution of extramedullary disease present before therapy.
  PR: normalization of peripheral counts and hepatosplenomegaly with bone marrow blasts reduced by 50% but >5% of cellularity except in cases of MDS/MPN with ≤ 5% blasts at baseline.
  Progression: ≥ 50% reduction from maximum response levels in granulocytes or platelets, and/or reduction in hemoglobin by ≥ 1.5 g/dL in the absence of another explanation; transfusion dependence.
Time Frame: Cycle 1 to disease progression or end of study, whichever occurred earlier (cycle length = 28 days). Median time on study was 4.1 months
Population: The full analysis set included all enrolled participants who received at least 1 dose of AMG 176.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
Participants
  Responders | 0 | 0
  Non-responders | 4 | 3

4. Secondary Outcome: Time to a Response According to the Uniform Response Criteria for MDS/MPN
Description: A responder was assessed as having CR or PR. CR: ≤ 5% myeloblasts with normal maturation of all cell lines and return to normal cellularity; osteomyelofibrosis was absent or equal to mild reticulin fibrosis; resolution of extramedullary disease present before therapy.
  PR: normalization of peripheral counts and hepatosplenomegaly with bone marrow blasts reduced by 50% but >5% of cellularity except in cases of MDS/MPN with ≤ 5% blasts at baseline.
Time Frame: as for outcome 3
Population: The full analysis set included all enrolled participants who received at least 1 dose of AMG 176. No participants were responders.
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response According to the Uniform Response Criteria for MDS/MPN
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 4
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Event-free Survival
Time Frame: as for outcome 3
Population: As pre-specified in Section 10 of the statistical analysis plan, EFS was not analyzed.
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of AMG 176
Description: AMG 176 plasma concentrations with values below the limit of quantification were set to zero. Pharmacokinetic (PK) parameters were determined from the time concentration profile using noncompartmental analysis.
Time Frame: Cycle 1: pre-dose, end of infusion (EOI), 3, 5, 7, 8, 24 hours post-infusion in weeks 1 and 2; pre-dose, EOI, 8 and 24 hours post-infusion in cycle 1 weeks 3 and 4
Population: The PK analysis set included all participants who received at least 1 dose of AMG 176 and had at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
ng/mL
  Cycle 1 day 1 | 18600 (16600) | 5650 (1790)
  Cycle 1 day 8 | 19500 (6600) | 14900 (5060)

8. Secondary Outcome: Time to Cmax (Tmax) of AMG 176
Description: AMG 176 plasma concentrations with values below the limit of quantification were set to zero. PK parameters were determined from the time concentration profile using noncompartmental analysis.
Time Frame: Cycle 1: pre-dose, EOI, 3, 5, 7, 8, 24 hours post-infusion in weeks 1 and 2; pre-dose, EOI, 8 and 24 hours post-infusion in cycle 1 weeks 3 and 4
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
hours
  Cycle 1 day 1 | 2.4 [2.2 to 5.3] | 2.5 [2.3 to 5.1]
  Cycle 1 day 8 | 2.5 [2.3 to 2.7] | 3.0 [2.3 to 3.1]

9. Secondary Outcome: Area Under the Plasma Concentration Time Curve From 0 to 168 Hours (AUC168hr) of AMG 176
Description: as for outcome 8
Time Frame: as for outcome 8
Population: The PK analysis set included all participants who received at least 1 dose of AMG 176 and had at least 1 PK sample collected. Participants with data available at each time point are included.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
hour*ng/mL
  Cycle 1 day 1 | 198000 (148000) | 75900 (32000)
  Cycle 1 day 8: number analyzed (Participants) | 3 | 3
  Cycle 1 day 8 | 167000 (146000) | 179000 (85600)

10. Secondary Outcome: Terminal Half-life of AMG 176
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
hours
  Cycle 1 day 1: number analyzed (Participants) | 4 | 2
  Cycle 1 day 1 | 27.0 [9.93 to 57.2] | 19.2 [10.4 to 27.9]
  Cycle 1 day 8: number analyzed (Participants) | 3 | 3
  Cycle 1 day 8 | 19.7 [5.10 to 40.8] | 21.1 [9.01 to 22.9]

11. Secondary Outcome: Clearance (CL) of AMG 176
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/hour/m^2
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
Number analyzed (Participants) | 4 | 3
mL/hour/m^2
  Cycle 1 day 1 | 1300 (1400) | 1890 (1070)
  Cycle 1 day 8: number analyzed (Participants) | 3 | 3
  Cycle 1 day 8 | 1150 (788) | 1540 (595)

ADVERSE EVENTS:
Time Frame: For all-cause mortality, from enrollment through end of study; median (min, max) time on study was 4.1 ( 2.2, 8.61) months. For serious and other AEs, from first dose of AMG 176 to up to 30 days after the last dose or end of study, whichever occurred first; median (min, max) duration was 2.7 ( 2.07, 4.73) months.
Arm/Group | Part 1A Dose Exploration: AMG 176 Dose Level 1 | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2
All-Cause Mortality (participants affected / at risk) | 3/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A Dose Exploration: AMG 176 Dose Level 1 (N=4) | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2 (N=3)
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Penile infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A Dose Exploration: AMG 176 Dose Level 1 (N=4) | Part 1A Dose Exploration: AMG 176 Dose Level 1 Then Dose Level 2 (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 0 | 1
Catheter site pruritus (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 3
Gait disturbance (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 1 | 0
Scrotal erythema (Reproductive system and breast disorders) | 1 | 0
Testicular haemorrhage (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was planned to be conducted in 3 parts and was discontinued early after the completion of Part 1A due to strategic reasons. No participants enrolled into Parts 1B and 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT05209152/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT05209152/SAP_001.pdf